CLINICAL TRIAL: NCT05824013
Title: Blood Caogulation Profile After Liver Resection. Comparison of Conventional Blood Coagulation Tests With Thromboelastography
Brief Title: Blood Coagulation Profile After Liver Resection.
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Sponsor
Other Study IDs: 5492
Record Dates: First submitted 2023-04-11; First posted 2023-04-21 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2023-04

CONDITIONS: Coagulation Disorder
MeSH Terms: conditions — Hemostatic Disorders | interventions — Thrombelastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: thromboelastography (TEG®6s) — blood samples for conventional coagulation test were obtained in vacutainer tubes from an arterial line. Two blood citrate samples (3 ml, sodium citrate solution, Vacuette® Blood Tubes) were also collected for the laboratory conventional coagulation tests (aPTT, INR, D-dimer levels, Antithrombin III) and TEG®6s assessment. The TEG parameters include reaction time (R), clot formation time (K), angle or α (K angle), maximum amplitude (MA), and amplitude at 30 minutes (LY30)

SUMMARY:
Liver resection is the treatment of choice in patients with primary or metastatic liver neoplasms, benign liver neoplasms and numerous biliary diseases. In these patients, in the postoperative period,several factors can induce a transient alteration of the synthesis hepatic coagulation factors such as size of the lesion liver, underlying liver disease (e.g. malignancy), pre-existing cirrhosis, duration of both surgery and vascular clamping, and blood loss. So far, some studies have shown that conventional coagulation tests indicate a hypocoagulable state which may lead to excessive transfusions of blood products or an increased risk of thromboembolic events related to delayed initiation of thromboprophylaxis in the postoperative period. In an attempt to optimizing the state of coagulation, recently there is increased interest for viscoelastic coagulation testing (thromboelastography and rotational thromboelastometry). The results of these studies have shown that these patients often have a hypercoagulable and non hypocoagulable profile as evidenced by conventional coagulation tests.

the purpose of the study is to evaluate whether the combination of coagulation tests conventional systems and new thromboelastography can increase the quality of surveillance of the coagulation state after liver surgery, in order to optimize the management of postoperative blood coagulation of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Elective liver resection surgery for liver cancer primary or metastatic
* Admission to surgical intensive care unit at the end of the surgery.

Exclusion Criteria:

* Renal disease (creatinine clearance < 30 ml/min)
* pregnancy
* Benign liver disease
* Emergency surgery
* Reintervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing liver surgery resective for primary or secondary neoplastic disease admitted to surgical intensive care unit at the end of surgery
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
blood coagulation profile | 12 hours
  Evaluate whether to use TEG®6s, in addition to coagulation tests conventional, optimizes the postoperative hemocoagulation management of patients undergoing resective liver surgery in terms of consumption transfusion of plasma and blood products.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, Italy

REFERENCES:
- [Result] Ardito F, Vellone M, Barbaro B, Grande G, Clemente G, Giovannini I, Federico B, Bonomo L, Nuzzo G, Giuliante F. Right and extended-right hepatectomies for unilobar colorectal metastases: impact of portal vein embolization on long-term outcome and liver recurrence. Surgery. 2013 Jun;153(6):801-10. doi: 10.1016/j.surg.2013.02.001. PMID 23701876
- [Result] Dumitrescu G, Januszkiewicz A, Agren A, Magnusson M, Isaksson B, Wernerman J. The temporal pattern of postoperative coagulation status in patients undergoing major liver surgery. Thromb Res. 2015 Aug;136(2):402-7. doi: 10.1016/j.thromres.2015.05.023. Epub 2015 May 24. PMID 26048400
- [Result] Blasi A, Molina V, Sanchez-Cabus S, Balust J, Garcia-Valdecasas JC, Taura P. Prediction of thromboembolic complications after liver resection for cholangiocarcinoma: is there a place for thromboelastometry? Blood Coagul Fibrinolysis. 2018 Jan;29(1):61-66. doi: 10.1097/MBC.0000000000000672. PMID 29045240